CLINICAL TRIAL: NCT05092178
Title: Effect of Calorie-restricted Diet and Exercise Intervention vs Exercise on the Knee Function of Metabolic Syndrome Patients With Degenerate Meniscus Lesions, a Randomized Controlled Study
Brief Title: Calorie Restricted Diet and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Hongyu Wang, Principal Investigator, Shenzhen People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: exercise01
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calorie restricted diet and exercise intervention (Experimental): The CR diet and exercise group received a balanced diet with an energy consists carbohydrates 45-65%; fat 20-35%; and protein 10- 35% and a deficit of 600 kcal/day from their daily energy requirement.
  The exercise intervention included aerobic exercises and resistance exercise, flexibility exercises about 150 minutes for ≥2 d/week for 6 months.
  Interventions: Behavioral: calorie restricted diet and exercise
- exercise group (Active Comparator): In exercise alone group, participants then underwent their usual habitual dietary diet and the above exercise intervention during the program.
  Interventions: Behavioral: exercise alone

INTERVENTIONS:
Behavioral: calorie restricted diet and exercise — The CR diet and exercise group received a balanced diet with an energy consists carbohydrates 45-65%; fat 20-35%; and protein 10- 35% and a deficit of 600 kcal/day from their daily energy requirement.The exercise intervention consists of aerobic exercises and resistance exercise, flexibility exercises about 150 minutes for≥2 d•wk for six months. The aerobic exercises included walking on a treadmill, stationary cycling for at least 30 minutes for≥2 d•wk, while, resistance exercises included nine upper-extremity and lower-extremity exercise with weighting lift machines for ≥2 d•wk, while, flexibility exercise including the major muscle-tendon groups (a total of 60 s per exercise) for ≥2 d•wk. Participants performed 1 or 2 sets with 8-12 repetitions of each exercise. The exercise sessions were monitored by telephone video.
  Arms: Calorie restricted diet and exercise intervention
Behavioral: exercise alone — In exercise alone group, participants then underwent their usual habitual dietary diet and the above exercise intervention during the program.
  Arms: exercise group

SUMMARY:
Calorie-restricted(CR) diet and exercise were effective to reduce Metabolic syndrome(MetS), however, its effect on knee functions for MetS patients with degenerate meniscus lesions(DMLs) was still poorly investigated.

DETAILED DESCRIPTION:
The CR diet and exercise group received a balanced diet with an energy consists carbohydrates 45-65%; fat 20-35%; and protein 10- 35% and a deficit of 600 kcal/day from their daily energy requirement. Total daily energy intake of 1200-2000 kcal/day were based on baseline weight, and for safety, no woman was provided with less than 1100 kcals/d and no man less than 1300 kcals/d. The energy of the intake calorie restricted diet per day was calculated based on the detailed composition of meals, such as rice, vegetables, eggs, pork, and beef, using the Chinese food composition tables. Our diets were cooked with traditional Chinese cooking methods such as boiling, stir-frying, and stewing. During the intervention, other lipid-lowering drugs were not allowed to intake supplement as it alters the outcome. Participants receive education or counseling by a dietitian for modulations of their caloric intake weekly.

The exercise intervention included aerobic exercises and resistance exercise, flexibility exercises about 150 minutes for ≥2 d/week for 6 months. The aerobic exercises included walking on a treadmill, stationary cycling for at least 30 minutes for≥2 d/week. Resistance exercises included nine upper-extremity and lower-extremity exercise with weighting lift machines for ≥2 d/week, while, flexibility exercise including the major muscle-tendon groups (a total of 60 s per exercise) for ≥2 d/week. Participants performed 1 or 2 sets with 8-12 repetitions of each exercise. The exercise sessions were monitored by telephone video. Patients who complete at least 80% of diet restriction and exercise were included in analysis. Calorie restricted diet and exercise group contain both the above intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Must be age between 35 and 70 years old;

  * Clinical diagnosis of metabolic syndrome;

Exclusion Criteria:

* • Must be able to have no acute knee injury such as car crash or acute sports injury;

  * Must be able to have no knee surgeries history;
  * Must be able to have no rheumatoid arthritis or serious knee osteoarthritis with deformity;
  * Must be able to have no contraindications to MRI;
  * Must be able to have no severe cardiopulmonary disease;
  * Must be able to have no musculoskeletal or neuromuscular impairments ;
  * Must be able to have good visual, hearing, or cognitive;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
The Knee injury and Osteoarthritis Outcome Score (KOOS) score change | Change from Baseline KOOS at 6 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS) holds five subscales including: Pain (9 items); other Symptoms (7 items); Activities of Daily Living (ADL, 17 items); Sport and Recreation function (Sport/Rec, 5 items); and knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems)
The International Knee Documentation Committee Subjective Knee Evaluation score change | Change from Baseline IKDC at 6 months
  The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) score questionnaire contains 18 items (7 items for symptoms, 1 item for sport activity, 9 items for daily activities, and 1 item for current knee function.) The total score is transformed to a value on a scale of 0 to 100, with 100 representing the highest knee function and 0 is the worst.
The Knee injury and Osteoarthritis Outcome Score (KOOS) score change | Change from Baseline KOOS at 12 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS) holds five subscales including: Pain (9 items); other Symptoms (7 items); Activities of Daily Living (ADL, 17 items); Sport and Recreation function (Sport/Rec, 5 items); and knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems)
The International Knee Documentation Committee Subjective Knee Evaluation score change | Change from Baseline IKDC at 12 months
  The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) score questionnaire contains 18 items (7 items for symptoms, 1 item for sport activity, 9 items for daily activities, and 1 item for current knee function.) The total score is transformed to a value on a scale of 0 to 100, with 100 representing the highest knee function and 0 is the worst.

SECONDARY OUTCOMES:
subscales of KOOS pain score change | Change from Baseline pain at 6 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life.The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
subscales of KOOS pain score change | Change from Baseline pain at 12 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life.The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
subscales of KOOS symptoms score change | Change from Baseline symptoms at 6 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
subscales of KOOS symptoms score change | Change from Baseline symptoms at 12 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
KOOS activity of daily living change | Change from Baseline activity of daily living at 6 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
KOOS activity of daily living change | Change from Baseline activity of daily living at 12 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
sport and recreational function change | Change from Baseline sport and recreational function at 6 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
sport and recreational function change | Change from Baseline sport and recreational function at 12 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
knee related quality of life change | Change from Baseline knee related quality of life at 6 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
knee related quality of life change | Change from Baseline knee related quality of life at 12 months
  Secondary outcomes include five subscales of the KOOS covered pain, symptoms, activity of daily living, sport and recreational function, and knee related quality of life. The minimum is 0 points, the maximum is 4 points. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
systolic blood pressure change | Change from Baseline systolic blood pressure at 6 months
  systolic blood pressure /mmHg
systolic blood pressure change | Change from Baseline systolic blood pressure at 12 months
  systolic blood pressure /mmHg
diastolic blood pressure change | Change from Baseline diastolic blood pressure at 6 months
  diastolic blood pressure/mmHg
diastolic blood pressure change | Change from Baseline diastolic blood pressure at 12 months
  diastolic blood pressure/mmHg
body mass index change | Change from Baseline body mass index at 6 months
  body mass index /kg/㎡
body mass index change | Change from Baseline body mass index at 12 months
  body mass index /kg/㎡
weight change | Change from Baseline weight at 6 months
  Weight-kg
weight change | Change from Baseline weight at 12 months
  Weight-kg
high-density lipoprotein cholesterol change | Change from Baseline high-density lipoprotein cholesterol at 6 months
  high-density lipoprotein cholesterol (mmol/L)
high-density lipoprotein cholesterol change | Change from Baseline high-density lipoprotein cholesterol at 12 months
  high-density lipoprotein cholesterol (mmol/L)
low-density lipoprotein cholesterol change | Change from Baseline low-density lipoprotein cholesterol at 6 months
  low-density lipoprotein cholesterol (mmol/L)
low-density lipoprotein cholesterol change | Change from Baseline low-density lipoprotein cholesterol at 12 months
  low-density lipoprotein cholesterol (mmol/L)
triglycerides change | Change from Baseline triglycerides at 6 months
  triglycerides (mmol/l)
triglycerides change | Change from Baseline triglycerides at 12 months
  triglycerides (mmol/l)
total cholesterol change | Change from Baseline total cholesterol at 6 months
  total cholesterol (mmol/L)
total cholesterol change | Change from Baseline total cholesterol at 12 months
  total cholesterol (mmol/L)
fast blood glucose change | Change from Baseline fast blood glucose at 6 months
  fast blood glucose (mmol/L)
fast blood glucose change | Change from Baseline fast blood glucose at 12 months
  fast blood glucose (mmol/L)
waist circumstance change | Change from Baseline waist circumstance at 6 months
  waist circumstance (cm)
waist circumstance change | Change from Baseline waist circumstance at 12 months
  waist circumstance (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning, China